CLINICAL TRIAL: NCT03552016
Title: Evaluation of Progression of Myopia in Children Treated With Vitamin B2 and Outdoor Sunlight Exposure
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funds and move of all investigators to other institutions.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Mohannad Al-Samarraie, MD, Assistant Professor of Clinical Ophthalmology, Virginia Commonwealth University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011340 HS
Record Dates: First submitted 2018-05-28; First posted 2018-06-11 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Axial Myopia; Refractive Errors
Keywords: Myopia; Axial Myopia; Children; Refractive Error; Riboflavin; Vitamin B2
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Riboflavin

STUDY DESIGN:
Intervention Model Description: This is a 1:1:1 double-blinded randomized study for children ages 6-12 year old with axial myopia who will be treated with one of three different doses of oral riboflavin. Expected number of participants is 100.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The researchers involved, the project investigator, and the patients will be blinded from knowing which patient will get which treatment by assigning a number to each patient and having that patient take that number to the pharmacy where they will pick up their riboflavin. The dosage of riboflavin given to the patient will be chosen by the "number" that the patient gives to the pharmacy. There will be no labels revealing the dose of riboflavin that the patient receives. There will be placebo dose which contains a small dose of riboflavin that has been shown to not reach therapeutic levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 200 mg Riboflavin (oral) (Experimental): These patients (approximately 1/3rd of all patients enrolled in the study) will be given 200 mg oral riboflavin each day for 6 months and be encouraged to play outside for 30 minutes a day every day.
  Interventions: Drug: Oral Riboflavin
- 400 mg Riboflavin (oral) (Experimental): These patients (approximately 1/3rd of all patients enrolled in the study) will be given 400 mg oral riboflavin each day for 6 months and be encouraged to play outside for 30 minutes a day every day.
  Interventions: Drug: Oral Riboflavin
- 0 mg Riboflavin (oral) (Placebo Comparator): These patients (approximately 1/3rd of all patients enrolled in the study) will be given 0 mg oral riboflavin (placebo) each day for 6 months and be encouraged to play outside for 30 minutes a day every day.
  Interventions: Drug: Oral Riboflavin

INTERVENTIONS:
Drug: Oral Riboflavin — The intervention doses will be 200 mg oral riboflavin and 400 mg oral riboflavin doses; the placebo dose will be 0 mg of oral riboflavin
  Other Names: Vitamin B2

SUMMARY:
The investigators plan on using riboflavin (a Vitamin that can easily be taken orally each day) and having the children involved in the study play outside (where there is UV light created by the sun) in order to prevent the eye from becoming progressively more near-sighted.

DETAILED DESCRIPTION:
Myopia is equivalent to the colloquial term known as near-sightedness. This, in short, means that the image of one's environment is projected in front of the retina (rather than directly on the retina, which is ideal). Of course, glasses can be used to correct the image disparity that is created by being near-sighted (that is why a lot of people need glasses for blurry vision). However, glasses and spectacles and contacts do not correct the underlying problem. Most near-sightedness is due to the eye being "too long" and therefore the image projects in front of the retina. Ideally, if we could prevent the eye from becoming abnormally "long", then we could prevent the progression of near-sightedness. Indeed, a child may only be slightly near-sighted early in life, but as he/she continues to perform activities within an arms length of their environment, they can become progressively near-sighted. Besides spectacle correction, people have tried topical atropine drops (medicated eye drops) and rigid contact lenses (orthokeratology) to attempt to correct near-sightedness. Atropine drops take a lot of cooperation from parent and child. Orthokeratology also requires a lot of cooperation, but also, does not permanently stall myopic progression. The investigators suggest a different means of potentially preventing near-sightedness from getting worse (and thus prevent the eye from getting "too long"). The investigators plan on using riboflavin (a Vitamin that can easily be taken orally each day) and having the children involved in the study play outside (where there is UV light created by the sun) in order to prevent the eye from becoming progressively more near-sighted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children ages 6-12 years old with myopia more than 0.50 D and astigmatism no more than 1.5 D.
* Caretakers who choose to enroll their child in the study must agree to participate in the study on their own will after knowledge of potential alternatives (spectacle correction, orthokeratology, atropine eye drops, etc.) are explained to the patient's caretaker.

Exclusion Criteria:

* Known allergy to riboflavin
* Birth history of premature birth
* Developmental delay or other neurological or mental conditions
* Major systemic health problems
* Significant anisometropia more than 1.5 Diopters
* Any other eye condition which may complicate interpretation of data including: congenital glaucoma, congenital cataract, ectatic corneal condition, amblyopia or strabismus.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2029-10-10 (Estimated); Study Completion 2030-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in cycloplegic refraction | 3 years
  We will measure the average change in cycloplegic refraction over 3 years in each treatment/study group.

SECONDARY OUTCOMES:
Change in axial length | 3 years
  Change in axial length over 3 years in each treatment/study group.
Change in keratometry values | 3 years
  Change in keratometry values over 3 years in each study group.
Change in uncorrected best visual acuity | 3 years
  Change in uncorrected best visual acuity over 3 years in each study group.

CONTACTS AND LOCATIONS:
Overall Officials: Mohannad Al-Samarraie, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No